CLINICAL TRIAL: NCT06962683
Title: Post-surgery Muscle Preservation Through Blood Flow Restriction Training in Orthopedic Spinal Surgery
Brief Title: Post-surgery Muscle Preservation and Pain Reduction Through Blood Flow Restriction Training in Orthopedic Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBonn_WBS_BFR
Record Dates: First submitted 2025-04-15; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Muscle Atrophy; Postoperative Pain; Spondylolisthesis; Spondylodiskitis
MeSH Terms: conditions — Muscular Atrophy; Pain, Postoperative; Spondylolisthesis; Discitis | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): The first group will serve as the control group and will receive an additional daily Sham BFR intervention of 20mmHg postoperatively as part of routine clinical care.
  Interventions: Other: Sham-BFR
- Intervention Group (Experimental): The second group will serve as the intervention group and will receive an additional daily passiveBFR intervention with 80% of the individual LOP postoperatively as part of routine clinical care.
  Interventions: Other: Blood-Flow-Restriction Training

INTERVENTIONS:
Other: Blood-Flow-Restriction Training — For the pBFR intervention, the Personalized Tourniquet System for Blood Flow Restriction from Delfi Medical Innovations Inc. (Vancouver, Canada) were used. The cuffs were applied to both lower extremities as far proximally as possible and were connected to the control device. Before starting the training program, the individual LOP was measured of both lower limb in a restring, laying position by the control device. The Intervention-Group performed the training at 80% of their individual LOP. The training was performed alternately on both lower extremities. The time intervals were set at five minutes occlusion and five minutes rest. Each leg received five intervals of BFR-induced occlusion training, resulting in a total 50 minutes of daily training. During the entire training period, the patient was in a resting position, laying in the hospital bed.
  Other Names: BFR
  Arms: Intervention Group
Other: Sham-BFR — For the sham-BFR intervention, the Personalized Tourniquet System for Blood Flow Restriction from Delfi Medical Innovations Inc. (Vancouver, Canada) were used. The cuffs were applied to both lower extremities as far proximally as possible and were connected to the control device. Before starting the training program, the individual LOP was measured of both lower limb in a restring, laying position by the control device. The Control-Group was trained with a fixed pressure of 20 mmHg, independent of their individual LOP. The training was performed alternately on both lower extremities. The time intervals were set at five minutes occlusion and five minutes rest. Each leg received five intervals of BFR-induced occlusion training, resulting in a total 50 minutes of daily training. During the entire training period, the patient was in a resting position, laying in the hospital bed.
  Arms: Control Group

SUMMARY:
This project investigates the effects of the Blood-Flow-Restriction (BFR) training method on postoperative muscle atrophy and pain after spinal surgery. Two groups are formed for this purpose. The intervention group receives a everyday BFR training during the postoperative stay at an individually measured occlusion pressure of 60-80%. The control group performs sham-BFR training at a fixed occlusion pressure of 20mmHg. The examinations are carried out before and several times after the operation (longest follow-up: 6 months). Among other things, muscle mass, muscle strength, pain perception and quality of life are assessed using questionnaires.

DETAILED DESCRIPTION:
Methodology and implementation Type of study

Prospective, interventional study in the context of clinical orthopedic routine (Non-AMG, Non-MPG):

This scientific project investigates the influence of blood-flow restriction training as a therapeutic intervention after spinal surgery for postoperative muscle preservation.

Study design Parallel study design The aim of this study is to investigate the influence of postoperative blood-flow restriction (BFR) application on muscle preservation and muscular-functional rehabilitation after spinal surgery. Postoperative muscle mass and strength loss is related not only to the size of the surgical procedure, but also to the prolonged rehabilitation after spine surgery. Since our patients are not able to perform large mechanical loads for a longer period of time (usually six weeks), we use the BFR training method as a training intervention.

The thesis of this work focuses the postoperative use of BFR training to reduce muscle atrophy during hospitalisation phase, and the supporting effects of BFR-Training on functional rehabilitation. For this purpose, a partially blinded randomised controlled trial will treat one group with BFR and one group with Sham-BFR and compare the results.

Classification of patients and study procedure Subjects who fulfil the above-mentioned inclusion criteria for study participation will be informed orally and by means of an information sheet about the planned study by the investigator and given written information.

Prior to the start of the study, the written consent of the subjects to participate in the study will be obtained. The study takes into account the ethical principles of the Declaration of Helsinki in its current version (2013).

Randomisation of patients The patients will be divided into two groups of 25 patients each. Randomisation will be done by classical analogue double lottery.

1. Control (CG) The first group will serve as the control group and will receive an additional daily Sham BFR intervention of 20mmHg postoperatively as part of routine clinical care.
2. BFR intervention (BFR) The second group serves as the intervention group and receives an additional daily BFR intervention of 60-80% of the individual arterial occlusion pressure postoperatively as part of routine clinical care.

Description of the interventions Intervention: Blood-Flow Restriction Training (BFR). BFR training involves the application of tourniquets during a passive or active movement intervention to provide an additive metabolic stimulus. The tourniquets are applied as far as possible proximally to the thigh and a pressure is applied during the movement that suppresses only part of the venous return of an extremity (=venous pooling). Venous occlusion is induced by a cuff system routinely used in strength training (Delfi Medical Innovations Inc., Vancouver, Canada). The pressure applied is calculated on the basis of the individual occlusion pressure via duplex sonography at the start of each training session. The test person lies at rest while the cuff is inflated until no more blood flow can be detected in the extremity (= occlusion pressure). Of this occlusion pressure, 60-80% is subsequently used for the BFR intervention. The loading protocol provides for daily units of 60 minutes at intervals (5 minutes occlusion + 5 minutes free flow, six times in total), over a period of two to 14 days.

Control: Control group, Sham-BFR (CG). Patients in the control group (CG) perform the same exercise protocol as patients in the BFR intervention group, except that they receive the standardized low BFR pressure of 20mmHg.

Investigation/aim parameters of the study Investigations For the purpose of this project, the examinations will be divided into basal examinations and in-rehabilitation examinations.

1. Basal examinations All participating patients will undergo a multi-layered battery of tests before and after surgery, as well as long-term post-operative follow-up at 3, 6 and 12 months. The basal examinations take place on the premises of the orthopaedic clinic of the University Hospital Bonn. Examinations include measurement of muscle mass, muscle strength, pain perception and subjective questionnaires.
2. In-rehabilitation monitoring Vital signs such as blood pressure, pulse, oxygen saturation are taken before and after exercise with BFR, and a capillary blood sample is taken to show venous blood gases.

Study population

Patient inclusion criteria:

* The study includes all patients with a medical indication for spinal surgical therapy (including herniated disc, vertebral fracture, spinal stenosis, spondylodiscitis, etc).
* All participating patients have given their written informed consent to participate in the study.
* Patients aged between 18-85 years will be included.

Patient exclusion criteria:

* Acute or chronic infections of the extremities.
* Pregnancy and lactation
* Inability to undergo surgery

Number of patients: 50 (two groups with 25 subjects each)

Discontinuation of the study in one patient (drop-out)

One or more of the following circumstances may lead to a patient dropping out of the study (this patient will be counted as a drop-out):

* Withdrawal of the patient's consent without giving a reason.
* Occurrence of an exclusion criterion
* Violation of the study protocol
* Participation in < 80% of the intervention sessions

Statistical calculation of the number of cases A power analysis performed using G*Power 3.1.9. assuming a mean effect size (f) of 0.25, an alpha error of 0.05 and a test power of (1-β) of 0.85 for the analysis of variance with repeated measures resulted in an optimal sample size of N = 26 (i.e. 13 subjects per group).

Because of the long follow-up period of 6 months and the resulting increased possibility of drop-out patients, we agreed on a number of 25 subjects per group.

Recruitment measures The patients will be recruited from the patient pool of the Department of Orthopaedics and Trauma Surgery of the University Hospital Bonn.

Archiving and data protection All data generated in the course of the study are protected by data protection laws. Personal data will not be passed on or made accessible to the public by the medically responsible study director or the investigator (Alexander Franz) or any other person involved in the conduct of the study. Only pseudonymized patient data will be passed on and stored. The pseudonymization is carried out by means of an ascending numerical series by the medically responsible study director or the investigator. Only the investigators are allowed to assign the personal data to the study data. The allocation key is stored on an external hard drive and is managed by the principal investigator (Alexander Franz). After completion of the study, the allocation key is deleted and the data management is changed from pseudonymization to anonymization. The evaluation of the data will be anonymized. All data will be managed in accordance with data protection regulations.

ELIGIBILITY:
Inclusion Criteria:

* The study includes all patients with a medical indication for spinal surgical therapy (including herniated disc, vertebral fracture, spinal stenosis, spondylodiscitis, etc).
* All participating patients have given their written informed consent to participate in the study.
* Patients aged between 18-85 years will be included.

Exclusion Criteria:

* Acute or chronic infections of the extremities.
* Pregnancy and lactation
* Inability to undergo surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Muscle Mass | Pre- to 6 weeks Post Surgery
  BIA-/ DXA-Measurement

SECONDARY OUTCOMES:
Perceived Pain | Pre- to 6 weeks Post Surgery
  VAS 100mm

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No